CLINICAL TRIAL: NCT05008172
Title: Observation vs Embolization in Severe Splenic Injury: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Thomas Carver, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00040687
Record Dates: First submitted 2021-04-22; First posted 2021-08-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2023-11

CONDITIONS: Spleen Injury
Keywords: Blunt Splenic Injury; Nonoperative management; Splenic artery embolization

STUDY DESIGN:
Intervention Model Description: Once the attending surgeon decides on NOM the patient will be approached for enrollment by the ED Resuscitation Team. Randomization to prophylactic SAE vs observation will occur in block fashion.
Masking Description: Due to the interventional nature of this study (embolization vs observation), it will not be possible to mask providers or participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Splenic Artery Embolization (SAE) (Experimental): If a patient is randomized to the SAE arm, the Interventional Radiology (IR) team will be notified of the patient's enrollment. The timing of embolization is left to the IR team but will occur within 6-12 hours of enrollment.
  Interventions: Procedure: Splenic Artery Embolization
- Observation (No Intervention): Patients assigned to the observation arm will be transferred from the trauma bay to floor or the ICU for monitoring and continuous care under the Trauma team.

INTERVENTIONS:
Procedure: Splenic Artery Embolization — The decision for proximal or distal (selective) embolization is at the discretion of the Interventional Radiologist. For patients with angiographically evident injury, the choice of embolization site will be left to the discretion of the operator. For patients without angiographically evident injury, proximal splenic embolization will be performed with approved materials (coils or plugs for most patients) within the main splenic artery. The embolization endpoint will be hemostasis in the main splenic artery.
  Arms: Splenic Artery Embolization (SAE)

SUMMARY:
Nonoperative management (NOM) of blunt splenic injuries has been the standard of care for decades. While many splenic injuries can be successfully observed, studies have demonstrated increased failure rates for higher grade injuries, which prompted some institutions to perform SAE prophylactically. The current literature comparing observation and SAE is limited to observational data and is frequently inconsistent. As such, the standard of care varies across institutions and both strategies are considered acceptable management for splenic injuries. Our own institution does not routinely perform SAE and our splenic salvage rate exceed 90% but the investigators noted an increased rate of NOM failure in patients with a contrast blush on CT. Contrast blush is a known risk factor for NOM failure and has been cited as a reason to perform SAE, but even within this population no randomized trials have been performed to demonstrate if SAE improves outcomes. The purpose of this project is to provide definitive high-quality evidence for the effectiveness of SAE to decrease the rate of NOM failure in high grade splenic injuries.

DETAILED DESCRIPTION:
Background

The spleen is the most commonly injured organ in patients who sustain blunt abdominal trauma.[1] Splenic trauma management has evolved significantly over the past 40 years, with non-operative management (NOM) considered the standard of care due to the decrease in morbidity, shorter length of hospitalization, and preservation of splenic function.[2] There are several controversial topics in the management of blunt splenic injuries (BSI) but the utilization of splenic artery embolization (SAE) in NOM is perhaps the biggest one.[3] Proponents of SAE cite higher success rates for NOM and some have even advocated that it should always be used in the following situations: 1) presence of contrast ¨blush¨ or extravasation on CT or angiography, 2) AAST Grade 3 injuries associated with moderate amount of hemoperitoneum, or 3) Patients with AAST Grade 4-5 injuries.[4] These criteria have never been validated prospectively and are simply associated with a higher risk for NOM failure. Opponents to SAE cite that this invasive approach has no effect on successful observation and that it is associated with higher complication rates (splenic infarction, splenic abscess, puncture site issues) when compared to observation alone.[5-7] There is limited evidence to guide the decision regarding SAE vs observation in patients sustaining high-risk BSI. Numerous observational studies on the role of SAE in splenic injury management have been published but their findings are inconclusive and often contradictory.[8, 9] Considering the inconsistent evidence and the lack of any high-quality data to inform best practice, clinical equipoise is achieved and a randomized controlled trial comparing observation to SAE is justified. Data from our own institution has shown that the presence of a contrast blush is associated with a much higher NOM failure rate (unpublished data). Based off that finding the investigators hypothesize that prophylactic SAE will improve NOM success in patients with high-risk BSI.

The contemporary management of splenic injury

The contemporary management of BSI began in the mid-1980's when the surgeons began publishing their data on NOM of splenic trauma in children. The adult trauma surgeons subsequently began using this approach when CT technology allowed for identification and classification of solid organ injuries.[10] The American Association for Surgery of Trauma (AAST) developed and subsequently validated a splenic injury grading scale, which provided a standardized nomenclature for those treating patients with BSI.[11, 12] In addition, the AAST grade was shown to correlate with risk of NOM failure and also allowed institutions to benchmark their splenic salvage rates. With increased success in NOM there were subsequent improvements in other clinical outcomes including lower rates of blood transfusion and decreased length of stay.[13]

NOM does carry some risks, the most significant of which is delayed splenic rupture. Typically occurring within 72-hours, delayed splenic rupture is a potentially life-threatening event that usually requires splenectomy.[14] Failure of NOM also occurs because of persistent bleeding, an ongoing transfusion requirement, or worsening abdominal pain that prompts the surgeon to perform a splenectomy. Since the advent of NOM, researchers have worked to identify the risk factors associated with failure. Increasing age, amount of hemoperitoneum, grade of organ injury, and presence of contrast extravasation have all been associated with NOM failure.[14, 15] While none of these are absolute contraindications to NOM they are used by some institutions as criteria for which to use prophylactic SAE in an attempt to improve splenic salvage.[16] When employed in a prophylactic manner, the splenic artery is embolized, which decreases the amount of blood flowing to the injured areas within the spleen.[17] Splenic infarction is not inevitable since some perfusion occurs through collateral circulation and splenic immune function is maintained even after embolization.[18] Despite the potential benefit, prophylactic SAE has not been universally adopted. In a multi-center retrospective study, Lee et al noted that there was a wide variation of SAE utilization in Level 1 trauma centers, ranging from 5.1% to 33%.[19] This finding is not unexpected considering that, in 2012, only 30% of trauma centers had a written guideline for the management of splenic injury.[20] Despite these issues, NOM has been the standard of care for more than 30 years and currently >85% of patients undergo an attempt at NOM.[2] In a recent meta-analysis, the success rate of NOM is ~8.3% of all patients but the role of SAE in improving NOM success rates is still unclear.[21]

Evidence for and against SAE in splenic injury

Recognizing that contrast extravasation on CT was a potential factor associated with NOM failure, the surgeons at Shock Trauma in Maryland reported their initial experience with17 patients who were successfully managed with prophylactic SAE.[10] In 1995 they published a larger series of patients with contrast extravasation on CT scan. All patients underwent formal angiography and those with extravasation on angio underwent SAE.[22] In that paper, 87 of 90 (96.7%) patients had a negative angiography and were successfully managed with observation alone. Successful NOM was noted in 56 of 60 (93.3%) patients with a positive angio and subsequent SAE.[22] While these papers provided evidence that SAE could be helpful in the management of BSI patients they did not provide evidence that one technique was better than the other.

In one prospective multi-center observational study, Banerjee compared NOM splenic outcomes in high-SAE utilization centers vs low-utilization centers. Despite similar patient characteristics at presentation, the high SAE centers were noted to have a 50% lower rate of failure of NOM (3.5 vs 7.6%, respectively).[20] Several additional studies have shown that the addition of prophylactic SAE improves NOM success rates[4, 9, 23] but these are limited by their lack of randomization.

While there is an abundance of data supporting SAE, there are several studies questioning the role of embolization in splenic injury. Smith, et al reported their experience from 2000-2004 when 25% of their patients underwent SAE.[24] They noted a rather high overall NOM failure rate (14%) but an even higher failure rate in the SAE group (27%). In a similar paper from the same time period, Harbrecht and colleagues noted an insignificant difference in success of NOM in the SAE group vs observation group (80% vs 77.8%, respectively).[25] Duchesne, et al found that SAE was associated with increased rates of sepsis and ARDS when compared to a group of patients who underwent immediate splenectomy, which raises concerns about the technique itself and emphasizes the importance of patient selection.[7] The splenic injury outcomes trial (SPOT) from 2014 also calls into question the utility of SAE.[26] In this prospective observational multi-center trial, the investigators found no significant difference in splenectomy rates with or without SAE (2.5% vs 3.5%).[26] They further expanded on the resource utilization aspect of SAE and theorized that if embolization was employed in the 15,000 patients with high grade splenic injury (based off current data) only 274 spleens would be saved. Considering the cost and logistics of SAE, there may not be enough of a societal benefit to justify widespread adoption of this technique.[26] Given these concerns, the investigaors feel that the best way to answer this question is through a randomized controlled trial.

Splenic Blush on CT

The first publications regarding the importance of splenic contrast blush after trauma were published in the 1990's but these reports were sporadic and limited by small sample sizes.[27] In addition, trauma surgeons were still grappling with what to do in patients with a contrast blush and often erred on the side of some intervention (either splenectomy or SAE).[28] In 2001, Omert and colleagues reviewed their series of 324 patients with splenic injury. There was an 11% rate of splenic blush but they found that a blush was not associated with NOM failure.[28] Post et al (2013) found that observation had a similar rate of successful NOM when compared to SAE in low grade splenic injuries.[29] Conversely, Alarhayem and his group in San Antonio found that blush on CT correlated with NOM failure even if no contrast extravasation was noted on formal angiogram.[30] Most recently, Zarzaur explored the effect of a contrast blush in 200 patients from 17 trauma centers.[31] While SAE was used in 59% of people, the splenectomy rate was similar between the SAE group (6.8%) and the observation group (7.6%). This review demonstrated that a contrast blush is associated with a high risk for failure but that SAE may not actually mitigate that risk.[31]

Our own institutional data has shown that the presence of a blush correlated with a higher risk for NOM failure but this data is limited because of the retrospective nature. Our institution rarely employs SAE for blunt splenic injury. For this reason, the investigators feel that our institution is ideal to study the role of SAE in high-risk splenic injury.

Innovation

To date there has only been one randomized controlled trial comparing prophylactic SAE to observation (SAE as needed) in high-grade splenic injuries.[16] While they showed no difference in splenectomy rates between groups there was a significant difference in the rate of unplanned embolization (29.2% in the observation group vs 1.5% in the prophylactic SAE group). Another important detail is that this trial did not include patients with contrast extravasation or blush on CT. Our proposed study will include patients with a splenic blush because there is enough conflicting data in the literature to justify including this patient population.

References:

1. Peitzman, A.B. and J.D. Richardson, Surgical treatment of injuries to the solid abdominal organs: a 50-year perspective from the Journal of Trauma. J Trauma, 2010. 69(5): p. 1011-21.
2. Stassen, N.A., et al., Selective nonoperative management of blunt splenic injury: an Eastern Association for the Surgery of Trauma practice management guideline. J Trauma Acute Care Surg, 2012. 73(5 Suppl 4): p. S294-300.
3. Olthof, D.C., C.H. van der Vlies, and J.C. Goslings, Evidence-Based Management and Controversies in Blunt Splenic Trauma. Curr Trauma Rep, 2017. 3(1): p. 32-37.
4. Bhullar, I.S., et al., Selective angiographic embolization of blunt splenic traumatic injuries in adults decreases failure rate of nonoperative management. J Trauma Acute Care Surg, 2012. 72(5): p. 1127-34.
5. Bilello, J.F., et al., After the embo: predicting non-hemorrhagic indications for splenectomy after angioembolization in patients with blunt trauma. Trauma Surg Acute Care Open, 2018. 3(1): p. e000159.
6. Ekeh, A.P., et al., Complications arising from splenic artery embolization: a review of an 11-year experience. Am J Surg, 2013. 205(3): p. 250-4; discussion 254.
7. Duchesne, J.C., et al., Proximal splenic angioembolization does not improve outcomes in treating blunt splenic injuries compared with splenectomy: a cohort analysis. J Trauma, 2008. 65(6): p. 1346-51; discussion 1351-3.
8. Haan, J.M., et al., Nonoperative management of blunt splenic injury: a 5-year experience. J Trauma, 2005. 58(3): p. 492-8.
9. Miller, P.R., et al., Prospective trial of angiography and embolization for all grade III to V blunt splenic injuries: nonoperative management success rate is significantly improved. J Am Coll Surg, 2014. 218(4): p. 644-8.
10. Sclafani, S.J., et al., Blunt splenic injuries: nonsurgical treatment with CT, arteriography, and transcatheter arterial embolization of the splenic artery. Radiology, 1991. 181(1): p. 189-96.
11. Tinkoff, G., et al., American Association for the Surgery of Trauma Organ Injury Scale I: spleen, liver, and kidney, validation based on the National Trauma Data Bank. J Am Coll Surg, 2008. 207(5): p. 646-55.
12. Moore, E.E., et al., Organ injury scaling: spleen and liver (1994 revision). J Trauma, 1995. 38(3): p. 323-4.
13. Peitzman, A.B., et al., Blunt splenic injury in adults: Multi-institutional Study of the Eastern Association for the Surgery of Trauma. J Trauma, 2000. 49(2): p. 177-87; discussion 187-9.
14. McIntyre, L.K., M. Schiff, and G.J. Jurkovich, Failure of nonoperative management of splenic injuries: causes and consequences. Arch Surg, 2005. 140(6): p. 563-8; discussion 568-9.
15. Bhangu, A., et al., Meta-analysis of predictive factors and outcomes for failure of non-operative management of blunt splenic trauma. Injury, 2012. 43(9): p. 1337-46.
16. Arvieux, C., et al., Effect of Prophylactic Embolization on Patients With Blunt Trauma at High Risk of Splenectomy: A Randomized Clinical Trial. JAMA Surg, 2020.
17. Schnuriger, B., et al., Outcomes of proximal versus distal splenic artery embolization after trauma: a systematic review and meta-analysis. J Trauma, 2011. 70(1): p. 252-60.
18. Skattum, J., et al., Preserved splenic function after angioembolisation of high grade injury. Injury, 2012. 43(1): p. 62-6.
19. Lee, J.T., et al., American Society of Emergency Radiology Multicenter Blunt Splenic Trauma Study: CT and Clinical Findings. Radiology, 2021. 299(1): p. 122-130.
20. Banerjee, A., et al., Trauma center variation in splenic artery embolization and spleen salvage: a multicenter analysis. J Trauma Acute Care Surg, 2013. 75(1): p. 69-74; discussion 74-5.
21. Requarth, J.A., R.B. D'Agostino, Jr., and P.R. Miller, Nonoperative management of adult blunt splenic injury with and without splenic artery embolotherapy: a meta-analysis. J Trauma, 2011. 71(4): p. 898-903; discussion 903.
22. Sclafani, S.J.A., et al., Nonoperative Salvage of Computed Tomography-Diagnosed Splenic Injuries - Utilization of Angiography for Triage and Embolization for Hemostasis. Journal of Trauma-Injury Infection and Critical Care, 1995. 39(5): p. 818-827.
23. Sabe, A.A., et al., The effects of splenic artery embolization on nonoperative management of blunt splenic injury: a 16-year experience. J Trauma, 2009. 67(3): p. 565-72; discussion 571-2.
24. Smith, H.E., et al., Splenic artery embolization: Have we gone too far? J Trauma, 2006. 61(3): p. 541-4; discussion 545-6.
25. Harbrecht, B.G., et al., Angiography for blunt splenic trauma does not improve the success rate of nonoperative management. J Trauma, 2007. 63(1): p. 44-9.
26. Zarzaur, B.L., et al., The splenic injury outcomes trial: An American Association for the Surgery of Trauma multi-institutional study. J Trauma Acute Care Surg, 2015. 79(3): p. 335-42.
27. Schurr, M.J., et al., Management of blunt splenic trauma: computed tomographic contrast blush predicts failure of nonoperative management. J Trauma, 1995. 39(3): p. 507-12; discussion 512-3.
28. Omert, L.A., et al., Implications of the "contrast blush" finding on computed tomographic scan of the spleen in trauma. J Trauma, 2001. 51(2): p. 272-277.
29. Post, R., et al., Computed Tomography Blush and Splenic Injury: Does It Always Require Angioembolization? Am Surg, 2013. 73: p. 1089-1092.
30. Alarhayem, A.Q., et al., "Blush at first sight": significance of computed tomographic and angiographic discrepancy in patients with blunt abdominal trauma. Am J Surg, 2015. 210(6): p. 1104-10; discussion 1110-1.
31. Zarzaur, B.L., et al., Natural history of splenic vascular abnormalities after blunt injury: A Western Trauma Association multicenter trial. J Trauma Acute Care Surg, 2017. 83(6): p. 999-1005.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with blunt splenic injury.
2. Age ≥ 18 years old
3. AAST Grade 3 spleen injuries with significant hemoperitoneum (2 or more areas of hemoperitoneum)
4. AAST Grade 3 with the presence of contrast blush or pseudoaneurysm on contrast CT scan or angiography
5. AAST Grade 4 and 5 spleen injuries regardless of the presence of blush

Exclusion Criteria:

1. Hemodynamic instability on arrival at the hospital
2. Patients undergoing immediate surgical exploration for splenic or other intra-abdominal injuries
3. Patients with non-contrast CT scan of the abdomen
4. Patients undergoing angioembolization for other injuries
5. Patients with severe traumatic brain injury (GCS 8 or less)
6. Patients who are unable to give consent
7. Patients with contraindications for angioembolization (severe contrast allergy, chronic kidney disease (not on dialysis))
8. Pregnancy
9. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Failure of nonoperative management | 30 days
  Need for splenectomy
Failure of nonoperative management | 30 days
  Need for splenorrhaphy
Failure of nonoperative management | 30 days
  Unplanned SAE

SECONDARY OUTCOMES:
Complication rates | 30 days
  Complications will include mortality rates and hospitalization length of stay
Procedural complications for SAE Arm | 30 days
  Patients undergoing SAE will also be evaluated for technical and procedural success

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Carver, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No